CLINICAL TRIAL: NCT06292715
Title: A Single-Arm Clinical Study Evaluating Microwave Ablation of the Spleen Combined With Splenic Artery Occlusion for Secondary Hypersplenism Treatment
Brief Title: Microwave Ablation With Splenic Artery Occlusion for Secondary Hypersplenism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Microwave Ablation01
Record Dates: First submitted 2024-02-15; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Secondary Hypersplenism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- microwave ablation of the spleen combined with splenic artery occlusion (Experimental): The ablation puncture needle is percutaneously punctured into the spleen under ultrasound guidance, and the ablation method of one needle and multi-point method and needle insertion and pulling is mostly used
  Interventions: Procedure: microwave ablation of the spleen; Other: Splenic artery balloon implantation

INTERVENTIONS:
Procedure: microwave ablation of the spleen — Ultrasound-guided percutaneous puncture for splenic ablation treatment
Other: Splenic artery balloon implantation — Splenic artery balloon implantation

SUMMARY:
This study assesses the effectiveness of microwave ablation of the spleen in conjunction with splenic artery occlusion for treating secondary hypersplenism.

DETAILED DESCRIPTION:
This open-label, single-arm, single-center clinical trial investigates the combined approach of microwave ablation of the spleen and splenic artery occlusion for managing secondary hypersplenism.

ELIGIBILITY:
Inclusion Criteria:

* 1. written informed consent signed prior to enrolment 2. age > 18 years, both sexes 3.Patients with severe hypersplenism secondary to cirrhosis with clinical diagnosis, White blood cells <3×109/L, and/or platelet <50×109/L 4.Patients who have been repeatedly given drugs to raise white blood cells and platelets in clinical practice have poor effect 5.Mental problems such as clinical symptoms or anxiety in patients require interventional treatment for hypersplenism

Exclusion Criteria:

* Patients with any of the following are not eligible for enrollment in this study

  1. Coagulopathy or other blood disorders
  2. Recent use of anticoagulant drugs
  3. Severe hypertension and cardiac insufficiency
  4. Bone marrow aspiration results showed bone marrow suppression
  5. Combined with other spleen malignant diseases
  6. Severe skin infection at the puncture site
  7. Participated in other clinical studies within 2 months prior to the start of the study
  8. Patient or his/her authorized person is unwilling to sign a written informed consent form or unwilling to comply with the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Portal venous pressure | Up to 1 year
  Portal venous pressure
Hepatic artery blood flow velocity | Up to 1 year
  Hepatic artery blood flow velocity
Routine blood test | Up to 1 year
  Platelet count
Adverse Events | Up to 1 year
  Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: WEI LU, PhD, Principal Investigator — Tianjin Cancer Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No